CLINICAL TRIAL: NCT01142635
Title: The Appearance of Electromyography on the Anaesthesia Monitor.
Brief Title: Electromyographic (EMG) on the Anaesthesia Monitor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Arvi Yli-Hankala/Professor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R08197M; 2008-008129-31 (EudraCT Number)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Anaesthesia
Keywords: Electroencephalogram; Electromyogram; Entropy Index; Bispectral Index; Neuromuscular blockade; rocuronium; Propofol; Intubation
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rocuronium bromide — Rocuronium, iv, 0,6 mg/kg diluted with saline to double volume, bolus, single dose
  Other Names: Esmeron
Drug: Rocuronium bromide — Rocuronium, iv, single dose, single bolus, 1.2 mg/kg
  Other Names: Esmeron.

SUMMARY:
Intubation may induce electromyographic (EMG) activity, causing depth of anaesthesia monitors to show misleadingly high values. The investigators want to investigate whether this EMG activity can be visually seen on the anaesthesia monitor.

DETAILED DESCRIPTION:
Patients are anaesthetized with target controlled infusion of propofol. To facilitate intubation, the patients are randomized to receive rocuronium either 0,6 mg/kg or 1,2 mg/kg. BIS, Entropy and the biosignal collected with the Entropy strip are collected on a computer. The visible biosignal on the anaesthesia monitor is recorded with a video camera. BIS, Entropy, biosignal and video clip of the anaesthesia monitor will be analyzed in detail.

ELIGIBILITY:
Inclusion Criteria:

* females giving informed consent
* age range 18-65 years
* elective surgery: gynaecological
* general anaesthesia
* ASA classification 1 or 2

Exclusion Criteria:

* pregnancy
* body mass index > 30
* disease affecting CNS
* overuse of alcohol
* drug abuse
* unability to understand, read or use Finnish language

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The behaviour of biosignal on the anaesthesia monitor | 30 minutes
  The visibility of elctromyogram and elctroencephalogram on the anaesthesia monitor

SECONDARY OUTCOMES:
The behaviour of depth of anaesthesia indexes (BIS, SE, RE) during intubation | 30 min
  Intubation-associated changes in the numerical values of BIS, SE, RE

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, MD, Study Chair — Tampere University Hospital; Arvi Yli-Hankala, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland